CLINICAL TRIAL: NCT01062386
Title: The Epidemiology of Malaria Among Children Under Five in Mbarara District, Uganda - A Cross-sectional Population-based Survey 2010
Brief Title: Malaria Survey in Mbarara District, Uganda 2010
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Carolyn Nabasumba, Epicentre
Other Study IDs: Epicentre/Mba/2010/MalPrev
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Malaria
Keywords: prevalence; transmission; knowledge; attitude; practice
MeSH Terms: conditions — Malaria; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample for:
  Malaria rapid diagnostic test, Malaria Blood smear, Malaria PCR, Anopheles mosquitoes anti-saliva antibodies
Oversight: Data Monitoring Committee: No

SUMMARY:
Malaria is one of the major public health problems in Sub-Saharan Africa. In response to this threat, Roll Back Malaria (RBM) has rolled back a strategy using ACT as first line therapy for malaria episode, a wide distribution of Insecticide Treated Bednet (ITN), intermittent presumptive treatment of pregnant women and indoor residual spraying. Recent epidemiological observations suggested a decline in malaria prevalence in some countries but further evidences are still needed to confirm this evolution. The RBM strategy requires the use of reliable rapid diagnostic test (RDT) for which an operational assessment is necessary. Lastly, home-based management of malaria is also an important compound of this strategy. However, a better understanding of the actual use of antimalarial drugs, of the use of bednet and of the barrier to the use of health care is important to implement good quality strategies for malaria control.

This study is a cross-sectional community based survey made of two rounds (one in January 2010 and the second in June 2010). The general objective is to measure the prevalence of infection with Plasmodium falciparum at two periods of the year (at the moment of lowest and highest transmission based on the seasonal rainfalls) and to compare it with the prevalence estimated in 2004 after the rainy season for the same area. Specific objective are the estimation of the prevalence by age stratum, the analysis of the geographical distribution of the infection, the description of the parasitological characteristics, the assessment of three RDT, the description and the analysis of the prevention and care seek behaviours related to malaria.

The study area is the great Mbarara district located in south-west of Uganda. A three-stage cluster sampling method will be used. Spatial information will be collected with global positioning system and imported to Geographical Information System. Behaviour information will be collected through face to face interview.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Ages 1 month to 59 months

Exclusion Criteria:

* None

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children living in Great Mbarara district
Sampling Method: Probability Sample
Enrollment: 2320 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Proportion of malaria infections in children under 5 years of age | January-February 2010

SECONDARY OUTCOMES:
Proportion of families with knowledge, attitude and practice regarding malaria prevention | January-February 2010

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Nabasumba, Principal Investigator — Epicentre
Locations (1):
- Greater Mbarara district, Mbarara, Mbarara, Uganda